CLINICAL TRIAL: NCT02845167
Title: The Effect of Preoperative Exercise on Postoperative Outcome in AAA Patients: Pilot Study
Brief Title: Effect of Preoperative Exercise on Postoperative Outcome in AAA Patients: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medway NHS Foundation Trust (Other)
Collaborators: University of Kent (Other)
Responsible Party: Principal Investigator, Katharine Richardson, Dr Katharine Richardson, Medway NHS Foundation Trust
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 11/LO/1472
Record Dates: First submitted 2016-07-17; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Aortic Aneurysm, Abdominal; Surgery
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual-care only (No Intervention): Patients will receive usual-care only during the preoperative period.
- Preoperative exercise (Experimental): Patients will perform 3 consecutive days of 60 min submaximal cycling exercise at a moderate exercise intensity. During the 60 min of exercise, patients will be provided with three equally spaced 3min rest periods.
  Interventions: Other: Preoperative exercise

INTERVENTIONS:
Other: Preoperative exercise — Patients will perform 3 consecutive days of 60 min submaximal cycling exercise at a moderate exercise intensity. During the 60 min of exercise, patients will be provided with three equally spaced 3min rest periods
  Arms: Preoperative exercise

SUMMARY:
Basic animal research has demonstrated that exercise training can protect the myocardium from ischemia-reperfusion injury through several biological mechanisms . This effect of exercise training may be beneficial in the perioperative period when cardiac complications may arise. However, exercise induced cardioprotection is lost completely within 18 days of stopping the training program. This finding from animal research will be used to test the hypothesis that 3 days of consecutive exercise with the last bout conducted within the last 24/48 hours prior to surgery, will have a cardioprotective effect . Specifically, exercise has been shown to protect cardiac myocytes against reperfusion induced oxidative stress and mitochondria against reperfusion induced damage. This exercise mediated cardioprotection is observed in short moderate duration ischemia (i.e. 5-20 min) and moderate to severe (i.e.20-60 min) ischemic insults. The effects of exercise induced cardioprotection have only been investigated at cell level and it has not been shown whether this will translate into a reduction in postsurgical reperfusion injury and associated complications. To study this potential cardioprotective effect the investigators will aim to recruit patients who have a high risk of receiving reperfusion injury during surgery. Specifically, the investigators will recruit abdominal aortic aneurysm patients where the risk of heart complications is high. There is also currently no evidence in the published literature with regard to the effect of preoperative supervised exercise.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years of age.
* Patients able to give informed consent.
* Able to comply with the study protocol
* Patients undergoing open repair for an asymptomatic perirenal and infrarenal abdominal aortic aneurysm

Exclusion Criteria:

* Patients with severe disabling disorders limiting mobility, e.g. severe osteoarthritis
* Patients undergoing thoracoabdominal aneurysm surgery
* Patients physically unable or unwilling to undertake maximal cardiopulmonary exercise testing and the other fitness tests
* Patients younger than 18 years of age.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Length of in-hospital stay | Through study completion, on average up to 60 days post-surgery

SECONDARY OUTCOMES:
Postoperative mortality | 60 day mortality
Postoperative in-hospital complications | On average up to 5 days post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Richardson, Principal Investigator — Medway Maritime NHS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Powers SK, Quindry JC, Kavazis AN. Exercise-induced cardioprotection against myocardial ischemia-reperfusion injury. Free Radic Biol Med. 2008 Jan 15;44(2):193-201. doi: 10.1016/j.freeradbiomed.2007.02.006. Epub 2007 Feb 21. PMID 18191755
- [Background] Goldman L. Cardiac risks and complications of noncardiac surgery. Ann Intern Med. 1983 Apr;98(4):504-13. doi: 10.7326/0003-4819-98-4-504. PMID 6340579
- [Background] Lennon SL, Quindry JC, French JP, Kim S, Mehta JL, Powers SK. Exercise and myocardial tolerance to ischaemia-reperfusion. Acta Physiol Scand. 2004 Oct;182(2):161-9. doi: 10.1111/j.1365-201X.2004.01346.x. PMID 15450112
- [Background] Demirel HA, Powers SK, Zergeroglu MA, Shanely RA, Hamilton K, Coombes J, Naito H. Short-term exercise improves myocardial tolerance to in vivo ischemia-reperfusion in the rat. J Appl Physiol (1985). 2001 Nov;91(5):2205-12. doi: 10.1152/jappl.2001.91.5.2205. PMID 11641363
- [Background] Ascensao A, Ferreira R, Magalhaes J. Exercise-induced cardioprotection--biochemical, morphological and functional evidence in whole tissue and isolated mitochondria. Int J Cardiol. 2007 Apr 12;117(1):16-30. doi: 10.1016/j.ijcard.2006.04.076. Epub 2006 Jul 24. PMID 16860886
- [Background] Lennon SL, Quindry J, Hamilton KL, French J, Staib J, Mehta JL, Powers SK. Loss of exercise-induced cardioprotection after cessation of exercise. J Appl Physiol (1985). 2004 Apr;96(4):1299-305. doi: 10.1152/japplphysiol.00920.2003. Epub 2003 Dec 12. PMID 14672968